CLINICAL TRIAL: NCT02383810
Title: Randomized, Double-blind, Parallel Group, Placebo-controlled, Dose Finding Study in Colorectal Cancer Patients Receiving 5-FU-based Chemotherapy to Assess the Efficacy of Different Doses of s.c. Elsiglutide in the Prevention of Chemotherapy Induced Diarrhea (CID)
Brief Title: Dose Finding Study in Colorectal Cancer Patients Receiving 5-FU-based Chemotherapy to Assess the Efficacy of Elsiglutide in the Prevention of Chemotherapy Induced Diarrhea (CID)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Collaborators: Chiltern International Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TIDE-13-22
Record Dates: First submitted 2015-02-24; First posted 2015-03-09 (Estimated); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Drug and/or Toxin-induced Diarrhea
Keywords: Chemotherapy Induced Diarrhea (CID)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Elsiglutide 10 mg - target population (Active Comparator): Elsiglutide 10 mg once daily as s.c. injection for 4 consecutive days in patients receiving 5-FU based chemotherapy
  Interventions: Drug: Elsiglutide
- Elsiglutide 20 mg - target population (Active Comparator): Elsiglutide 20 mg once daily as s.c. injection for 4 consecutive days in patients receiving F-FU based chemotherapy
  Interventions: Drug: Elsiglutide
- Elsiglutide 40 mg - target population (Active Comparator): Elsiglutide 40 mg once daily as s.c. injection for 4 consecutive days in patients receiving 5-FU based chemotherapy
  Interventions: Drug: Elsiglutide
- Placebo - target population (Placebo Comparator): Placebo once daily as s.c. injection for 4 consecutive days in patients receiving 5-FU based chemotherapy
  Interventions: Drug: Placebo
- Elsiglutide 10 mg - additional population (Active Comparator): Elsiglutide 10 mg once daily as s.c. injection for 4 consecutive days in patients receiving 5-FU based chemotherapy with monoclonal antibody.
  Interventions: Drug: Elsiglutide
- Elsiglutide 20 mg - additional population (Active Comparator): Elsiglutide 20 mg once daily as s.c. injection for 4 consecutive days in patients receiving 5-FU based chemotherapy with monoclonal antibody.
  Interventions: Drug: Elsiglutide
- Elsiglutide 40 mg - additional population (Active Comparator): Elsiglutide 40 mg once daily as s.c. injection for 4 consecutive days in patients receiving 5-FU based chemotherapy with monoclonal antibody.
  Interventions: Drug: Elsiglutide
- Placebo - additional population (Placebo Comparator): Placebo once daily as s.c. injection for 4 consecutive days in patients receiving 5-FU based chemotherapy with monoclonal antibody.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Elsiglutide
  Arms: Elsiglutide 10 mg - additional population; Elsiglutide 10 mg - target population; Elsiglutide 20 mg - additional population; Elsiglutide 20 mg - target population; Elsiglutide 40 mg - additional population; Elsiglutide 40 mg - target population
Drug: Placebo
  Arms: Placebo - additional population; Placebo - target population

SUMMARY:
This is a randomized, stratified, double-blind, double-dummy, parallel group, placebo-controlled, dose finding, multicentre, multinational, phase II study in patient with colorectal cancer receiving 5- Fluorouracil (5-FU)-based chemotherapy (FOLFOX or FOLFIRI). Patients will receive, starting from the day of chemotherapy administration, a single daily dose subcutaneously (s.c.) of elsiglutide 10, 20 or 40 mg or placebo for 4 consecutive days. Each patient will be in the study for 3 consecutive chemotherapy cycles. The treatment period for each patient will be 4 consecutive days at each of the first 2 chemotherapy cycles.

The primary objective is to compare the efficacy of 3 s.c. doses of elsiglutide versus (vs.) placebo and vs. each other dose in the prevention of CID in colorectal cancer patients treated with 5-FU based chemotherapy (FOLFOX or FOLFIRI) with no addition of a monoclonal antibody.

DETAILED DESCRIPTION:
This is a randomized, stratified, double-blind, double-dummy, parallel group, placebo-controlled, dose finding, multicentre, multinational, phase II study in patient with colorectal cancer receiving 5- Fluorouracil (5-FU)-based chemotherapy (FOLFOX -FOLinic acid, Fluorouracil, OXaliplatin chemotherapy regimen - or FOLFIRI - FOLinic acid, Fluorouracil, IRInotecan chemotherapy regimen). Patients will receive, starting from the day of chemotherapy administration, a single daily dose subcutaneously (s.c.) of elsiglutide 10, 20 or 40 mg or placebo for 4 consecutive days. Each patient will be in the study for 3 consecutive chemotherapy cycles. The treatment period for each patient will be 4 consecutive days at each of the first 2 chemotherapy cycles.

Randomization will be performed with a 1:1:1:1 treatment allocation and will be stratified by chemotherapy regimen and country. Two populations are planned for this study.

The population receiving FOLFOX or FOLFIRI without monoclonal antibody is defined as the Target population, while the population concomitantly receiving monoclonal antibody is defined as the Additional population.

Randomization in Target and Additional population are handled independently.

Primary Objective:

To compare the efficacy of 3 s.c. doses of elsiglutide versus (vs.) placebo and vs. each other dose in the prevention of CID in colorectal cancer patients treated with 5-FU based chemotherapy (FOLFOX or FOLFIRI) with no addition of a monoclonal antibody.

Secondary Objectives:

* As a secondary objective, the efficacy of 3 s.c. doses of elsiglutide vs. placebo and vs. each other dose in the prevention of CID in colorectal cancer patients treated with 5-FU based chemotherapy (FOLFOX or FOLFIRI) given in combination with a monoclonal antibody will be explored.
* Safety and tolerability of the administered repeated doses of elsiglutide will be evaluated.

Additionally the following secondary objectives will be explored:

* The pharmacokinetics (PK) of elsiglutide, and its metabolites in each patient who consents to undergo an exposure assessment after the first administration and at steady state. The influence of possible demographic and therapeutic covariates on the PK parameters and their variability will also be investigated. The possible relationship between exposure of elsiglutide and its metabolites and efficacy measures in the target and overall population will be explored.
* The economic impact of the 3 doses of elsiglutide vs. placebo and each other dose in the treatment of CID.
* The impact on patient's QoL (quality of life) of the different dosages vs. placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Male or female > 18 years of age;
3. Histologically or cytologically confirmed diagnosis of colorectal cancer

   * Inclusion in the Target Population: Scheduled to receive at least 3 consecutive cycles of the same regimen of FOLFOX or FOLFIRI without monoclonal antibody;
   * Inclusion in the Additional Population: Scheduled to receive at least 3 consecutive cycles of the same regimen of FOLFOX or FOLFIRI in combination with monoclonal antibody;
4. A performance status of ≤ 2 according to the Eastern Cooperative Oncology Group (ECOG) scale;
5. Non-childbearing female patient or female patient of childbearing potential using reliable contraceptive measures and having negative pregnancy test before treatment administration;
6. Able to read, understand, follow the study procedure and complete patient diary.

Inclusion criteria will be checked during the screening visit. Inclusion criteria 4 and 6 will be re-checked as applicable on Day 1 of Cycle 1 and Cycle 2.

Exclusion Criteria:

1. Any investigational drugs within 30 days before enrollment or foreseen use of investigational agents during the study;
2. Treatment with chemotherapy of any type within 12 months before enrollment;
3. Patient with any type of ostomy (temporary ostomy should be closed at least 6 months prior to enrollment);
4. Patient who underwent total colectomy;
5. Patient who had abdominal-perineal resection or surgery leaving the patient without a functioning rectum;
6. Any radiotherapy to the abdomen or pelvis in the 6 months prior to enrollment;
7. Scheduled to receive radiotherapy to abdomen or pelvis during the study;
8. a) Exclusion from the Target population Scheduled to receive any concomitant chemotherapeutic agent, other than FOLFOX or FOLFIRI agents; any type of monoclonal antibodies;

8. b) Exclusion from the Additional population Scheduled to receive any concomitant chemotherapeutic agent, other than FOLFOX or FOLFIRI agents;

9. Any type of condition leading to diarrhea, including but not limited to inflammatory bowel diseases (e.g. ulcerative colitis and Crohn's disease), diarrhea of presumed or confirmed infectious origin and irritable bowel syndrome, celiac disease, lactose intolerance, pancreas, liver or diverticular disease, alcohol abuse;

10. History of chronic (≥ 30 consecutive days) use of laxatives;

11. Active and ongoing systemic infection;

12. Lactating woman;

13. History of hypersensitivity or allergies to drugs or compounds potentially related to this investigational drug class;

14. Previous exposure to Glucagon-like peptide-2 (GLP-2) or other compounds in this investigational drug class;

15. Patient who participated in a previous study with elsiglutide;

16. Patient with abnormalities in selected laboratory parameters, including:

* Aspartate aminotransferase (AST) ≥ 5 x upper limit of normal
* Alanine aminotransferase (ALT) ≥ 5 x upper limit of normal
* Bilirubin > 1.5 x upper limit of normal
* Creatinine > 2 mg/dL (177 μmol/L)
* Albumine < 2 g/dL (20 g/L)
* Neutrophils < 1.5 x109/L
* Platelet count < 100 x109/L ;

  17. Any illness or condition that, in the opinion of the investigator, may confound the results of the study or pose unwarranted risk in administering the investigational product to the patient;

  18. Any medical condition that precludes the administration of chemotherapy;

  19. Use of laxatives within 7 days prior to study Day 1;

  20. Use of antibiotics within 7 days prior to study Day 1;

  21. Any diarrhea in the 48 hours preceding study drug administration on Day 1;

  22. Major surgery within the previous 21 days before study Day 1;

  23. Use of anti-diarrheal agents and probiotics within the 48 hours prior to study drug administration on study Day 1.

Exclusion criteria 1 to 18 will be checked during the screening visit. Exclusion criteria 19 to 23 should be checked on Day 1 of Cycle 1. Exclusion criteria 7, 8, 9, 11 and 17 to 23 will be re-checked on Day 1 of Cycle 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- Belarus (5):
  - State Institution "Republic Scientific and Practical Center of oncology and medical radiology n.a.N.N.Alexandrov", Lyasny, Minsk Oblast
  - Healthcare Institution Brest Regional Oncologic Dispensary, Brest
  - Institution Gomel Regional Clinical Oncology Dispensary, Homyel
  - Healthcare Institution Minsk City Clinical Oncologic Dispensary, Minsk
  - Healthcare Institution Mogilev Regional Oncologic Dispensary, Mogilev
- Bulgaria (6):
  - Specialized Hospital for active treatment in oncology - Haskovo Ltd, Haskovo
  - ''Multifunctional Hospital for Active Treatment Central Onco Hospital" Ltd, Plovdiv
  - Complex Oncology Centre - Plovdiv Ltd, Plovdiv
  - Multifunctional Hospital for Active Treatment for Women's Health Nadezhda Ltd., Sofia
  - "Specialized Hospital for Active Treatment of Oncology Diseases - Sofia city" EOOD, Sofia
  - "Specialized Hospital for Active Treatment ofOncologal Diseases - Sofia District", Sofia
- Pardubicka krajska nemocnice a.s, Pardubice, Czechia
- Klinikum Neuperlach, München, Germany
- Hungary (8):
  - Semmelweis Egyetem, ÁOK I. Sz. Belgyógyászati Klinika, Onkológiai Részleg, Budapest
  - Országos Onkológiai Intézet "C" Belgyógyászati-Onkológiai és Klinikai Farmakológiai Osztály, Budapest
  - Uzsoki Utcai Kórház Onkoradiológia, Sugárterápia, ővárosi Onkoradiológiai Központ, Budapest
  - Debreceni Egyetem, OEC Onkológiai Tanszék, Debrecen
  - Somogy Megyei Kaposi Mór Oktató Kórház Klinikai Onkológiai Osztály, Kaposvár
  - Jósa András Oktatókórház Onkoradiológiai Osztály, Nyíregyháza
  - Szegedi Tudományegyetem, ÁOK, Szent-Györgyi Albert Klinikai Központ Onkoterápiás Klinika, Szeged
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház Onkológiai Osztály, Szolnok
- Poland (3):
  - Centrum Medyczne Malgorzata, Gmina Śrem
  - Centrum Medyczne MrukMed, Rzeszów
  - Wojewódzki Szpital Zespolony im. Rydygiera, Torun
- Russia (21):
  - State Budgetary Healthcare Institution of Republic of Mordovia "Republican Oncology Dispensary", Saransk, Respublika Mordoviya
  - State Budgetary Healthcare Institution "Volgograd Regional Oncology Dispensary", Volzhsky, Volgograd Oblast
  - State Budgetary Institution of Arkhangelsk Region "Arkhangelsk Clinical Oncology Dispensary", Arkhangelsk
  - Non-State Healthcare Institution "Railway Clinical Hospital at Chelyabinsk Station of Joint Stock Company "Russian Railways", Chelyabinsk
  - State Healthcare Institution "Kursk Regional Clinical Oncology Dispensary", Kursk
  - Federal State Budgetary Institution "Russian Oncology Scientific Centre named after N.N. Blokhin" of the Russian Academy of Medical Science, Moscow
  - State Budgetary Healthcare Institution "City Clinical Hospital #40" of the Healthcare Department of Moscow, Moscow
  - State Budgetary Healthcare Institution of Moscow "Moscow City Oncology Hospital #62" of Healthcare Department of Moscow, Moscow
  - State Budgetary Healthcare Institution of Nizhny Novgorod region "Clinical Diagnostic centre", Nizhny Novgorod
  - State Budgetary Healthcare Institution of Nizhniy Novgorod Region "Nizhniy Novgorod Regional Oncology Dispensary", Nizhny Novgorod
  - Budgetary Healthcare Institution of Omsk Region "Clinical Oncology Dispensary", Omsk
  - State Budgetary Healthcare Institution "Orenburg Regional Clinical Oncology Dispensary", Orenburg
  - Budgetary Healthcare Institution of Orel Region "Orel Oncology Dispensary", Oryol
  - State Budgetary Healthcare Institution of Perm Territory "Perm Territorial Oncology Dispensary", Perm
  - State Budgetary Healthcare Institution of Stavropol Territory "Pyatigorsk Oncology Dispensary", Pyatigorsk
  - State Budgetary Educational Institution of Higher Professional Education "First Saint Petersburg State Medical University named after Academician I.P. Pavlov", Saint Petersburg
  - State Healthcare Institution "City Hospital #9" (Saint Petersburg Theoretical & Practical Centre of Coloproctology), Saint Petersburg
  - Research Institute of Pulmonology of State Budgetary Educational Institution of Higher Professional Education "First Saint Petersburg State Medical University named after Academician I.P. Pavlov" of the Ministry of Healthcare of the Russian Federation, Saint Petersburg
  - State Budgetary Healthcare Institution "Saint Petersburg Clinical Theoretical & Practical Centre of Special Types of Medical Care (Oncology)", Saint Petersburg
  - State Budgetary Healthcare Institution "Samara Regional Clinical Oncology Dispensary" (Chemotherapy Unit #1), Samara
  - State Budgetary Healthcare Institution "Republican Clinical Oncology Dispensary", Ufa
- Ukraine (9):
  - Chernigiv medical and prophylactic establishment "Chernigiv regional oncological center", Chernihiv
  - Communal Institution "Chernivtsi Regional clinical oncology dispensary", Chernivtsi
  - Communal Institution Dnipropetrovsk City Multifunctional Clinical Hospital #4, Dnipropetrovsk
  - Ivano-Frankivsk Regional Oncological Center, Ivano-Frankivsk
  - Communal Institution Kharkiv Regional Clinical Oncology Center, Kharkiv
  - Municipal institution "Kirovograd Regional Oncology Center", Kropyvnytskyi
  - Regional Сommunal Institution Kryvyi Rig Oncology Dispensary, Kryvyi Rih
  - Kyiv City Clinical Oncological Center, Kyiv
  - Lviv State Oncological Regional Treatment and Preventive Center, Lviv

RESULTS

PARTICIPANT FLOW:
Groups:
- Elsiglutide 10 mg - Target Population: Elsiglutide 10 mg once daily as s.c. injection for 4 consecutive days in patients receiving 5-FU based chemotherapy
  Elsiglutide
- Elsiglutide 20 mg - Target Population: Elsiglutide 20 mg once daily as s.c. injection for 4 consecutive days in patients receiving F-FU based chemotherapy
  Elsiglutide
- Elsiglutide 40 mg - Target Population: Elsiglutide 40 mg once daily as s.c. injection for 4 consecutive days in patients receiving 5-FU based chemotherapy
  Elsiglutide
- Placebo - Target Population: Placebo once daily as s.c. injection for 4 consecutive days in patients receiving 5-FU based chemotherapy
  Placebo
- Elsiglutide 10 mg - Additional Population: Elsiglutide 10 mg once daily as s.c. injection for 4 consecutive days in patients receiving 5-FU based chemotherapy with monoclonal antibody.
  Elsiglutide
- Elsiglutide 20 mg - Additional Population: Elsiglutide 20 mg once daily as s.c. injection for 4 consecutive days in patients receiving 5-FU based chemotherapy with monoclonal antibody.
  Elsiglutide
- Elsiglutide 40 mg - Additional Population: Elsiglutide 40 mg once daily as s.c. injection for 4 consecutive days in patients receiving 5-FU based chemotherapy with monoclonal antibody.
  Elsiglutide
- Placebo - Additional Population: Placebo once daily as s.c. injection for 4 consecutive days in patients receiving 5-FU based chemotherapy with monoclonal antibody.
  Placebo
Period: Overall Study
Arm/Group | Elsiglutide 10 mg - Target Population | Elsiglutide 20 mg - Target Population | Elsiglutide 40 mg - Target Population | Placebo - Target Population | Elsiglutide 10 mg - Additional Population | Elsiglutide 20 mg - Additional Population | Elsiglutide 40 mg - Additional Population | Placebo - Additional Population
Started | 120 | 122 | 120 | 123 | 4 | 4 | 3 | 2
Completed | 117 | 114 | 113 | 112 | 4 | 3 | 2 | 2
Not Completed | 3 | 8 | 7 | 11 | 0 | 1 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 4 | 5 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — other | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — subject did not receive study treatment | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) was defined as all randomized patients who received at least 1 dose of study medication (elsiglutide or placebo) and (at least part of) the chemotherapy regimen in Cycle 1. The FAS Target set was defined as all patients from the Target population who were eligible for the FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | Elsiglutide 10 mg - Target Population | Elsiglutide 20 mg - Target Population | Elsiglutide 40 mg - Target Population | Placebo - Target Population | Elsiglutide 10 mg - Additional Population | Elsiglutide 20 mg - Additional Population | Elsiglutide 40 mg - Additional Population | Placebo - Additional Population | Total
Number analyzed (Participants) | 120 | 121 | 120 | 123 | 4 | 4 | 3 | 2 | 497
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (10.42) | 59.0 (10.84) | 60.6 (8.44) | 61.9 (9.57) | 62.0 (8.76) | 55.8 (12.53) | 57.7 (4.04) | 57.0 (7.07) | 61 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 62 | 51 | 59 | 3 | 1 | 2 | 0 | 232
  Male | 66 | 59 | 69 | 64 | 1 | 3 | 1 | 2 | 265
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 118 | 120 | 117 | 123 | 4 | 4 | 3 | 2 | 491
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Experiencing a Maximum Grade ≥ 2 Diarrhea During the First Cycle of Chemotherapy in the Target Population
Description: The endpoint of primary interest for efficacy was the proportion of patients within the Target population experiencing a maximum Grade ≥ 2 diarrhea in Cycle 1 (as assessed by the Investigator). For patient 8031362 who withdrew consent after 11 day in Cycle 1, Investigator assessments for the individual diarrhea events were missing. The data were imputed as Grade 0 for the primary endpoint, in line with the patient's eDiary data.
  Additional population is not included in primary endpoint evaluation.
Time Frame: 15 days
Population: FAS Target population, not including additional population
Measure: Number; unit: percentage of patients
Arm/Group | Elsiglutide 10 mg - Target Population | Elsiglutide 20 mg - Target Population | Elsiglutide 40 mg - Target Population | Placebo - Target Population
Number analyzed (Participants) | 120 | 121 | 120 | 123
percentage of patients
  With maximum Grade ≥ 2 diarrhea | 2.5 | 5.0 | 5.8 | 9.8
  With maximum Grade < 2 diarrhea | 97.5 | 95.0 | 94.2 | 90.2
Statistical Analysis 1: Comparison: Elsiglutide 10 mg - Target Population vs Elsiglutide 20 mg - Target Population vs Elsiglutide 40 mg - Target Population vs Placebo - Target Population; Overall null hypothesis: All elsiglutide dose groups had equal proportion of subjects with max Grade≥2 diarrhea and this was equal to the one in the placebo group. This includes 6 individual hypotheses (i.e., 3 to compare each dose group vs. placebo and 3 to compare dose groups vs. each other). Raw p-values from Chi square tests were corrected for multiplicity according to the Hommel's procedure. Each of 6 hypotheses was then evaluated based on corrected p-value at alpha 0.10 (two-sided); Test type: Superiority — The overall hypothesis system was represented by the following pool of partial hypothesis systems: Hok: πGi = πGj i = 1 to 3, and j = 2 to 4, and k = 1 to 6, and i ≠ j HAk: πGi ≠πGj i = 1 to 3, and j = 2 to 4, and k = 1 to 6, and i ≠ j where πG is the probability of absence of Grade ≥2 CID for the Group. Each Ho involved 2 groups; p < 0.1, Chi-squared — Overall alpha level 0.10 was maintained by correction for multiplicity according to Hommel's procedure

ADVERSE EVENTS:
Time Frame: AEs were collected from signature of Informed Consent until End of Trial visit (Day 14 after start of last cycle). Duration of collection was 7-8 weeks for each patient.
Description: The safety (SAF) set was defined as all treated patients. "Patients treated" was defined as any patient who received any study medication (elsiglutide or placebo) on at least 1 day. SAF Overall set was defined as all patients who were part of the SAF (either of SAF Target set or of SAF Additional set). Adverse events are reported for Cycles 1+2.
Groups:
- Elsiglutide 10 mg - Overall Set; Elsiglutide 20 mg - Overall; Elsiglutide 40 mg - Overall; Placebo - Overall: Adverse events occurring during Cycle 1 + 2 are reported. The safety (SAF) set was defined as all treated patients. "Patients treated" was defined as any patient who received any study medication (elsiglutide or placebo) on at least 1 day. The SAF Overall set was defined as all patients who were part of the SAF (either of SAF Target set or of SAF Additional set).
Arm/Group | Elsiglutide 10 mg - Overall Set | Elsiglutide 20 mg - Overall | Elsiglutide 40 mg - Overall | Placebo - Overall
All-Cause Mortality (participants affected / at risk) | 1/124 | 1/125 | 2/123 | 3/125
Serious Adverse Events (participants affected / at risk) | 2/124 | 4/125 | 3/123 | 6/125
Other Adverse Events (participants affected / at risk) | 71/124 | 68/125 | 73/123 | 72/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elsiglutide 10 mg - Overall Set (N=124) | Elsiglutide 20 mg - Overall (N=125) | Elsiglutide 40 mg - Overall (N=123) | Placebo - Overall (N=125)
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 2
Soft tissue inflammation (General disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Calculus urethral (Renal and urinary disorders) | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Elsiglutide 10 mg - Overall Set (N=124) | Elsiglutide 20 mg - Overall (N=125) | Elsiglutide 40 mg - Overall (N=123) | Placebo - Overall (N=125)
Anaemia (Blood and lymphatic system disorders) | 6 | 7 | 7 | 9
Leukopenia (Blood and lymphatic system disorders) | 6 | 10 | 6 | 12
Neutropenia (Blood and lymphatic system disorders) | 32 | 29 | 26 | 32
Asthenia (General disorders) | 9 | 8 | 7 | 7
Injection site erythema (General disorders) | 1 | 3 | 10 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 11 | 7 | 7
Nausea (Gastrointestinal disorders) | 21 | 17 | 15 | 17
Vomiting (Gastrointestinal disorders) | 1 | 3 | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No